CLINICAL TRIAL: NCT06056778
Title: The Prevalence Evaluation of Systemic Lupus Erythematosus in Russian Patients With Reproductive Issues (PRISMA)
Acronym: PRISMA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3461R00069
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus, reproductive issues
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will be a non-interventional prospective study. Assessment of parameters will be carried out as if the patient is treated in a real-life clinical setting. The patients should be enrolled into this project after evaluation of eligibility criteria by the investigator in clinical sites who have an experience in management of patients with SLE. No additional procedures besides those already used in the routine clinical practice will be applied to the patients.

The purpose of this study is to estimate prevalence of confirmed SLE in patients in rheumatological settings who has the reproductive issues and certain clinical and laboratory manifestations specific for immunoinflammatory diseases in Russia.

We will follow all the local regulatory requirements regarding adverse event reporting (pharmacovigilance).

It is planned to enrol 2000 patients in clinical sites in Russian Federation (N ≤ 15).

The study will include two visits. During the screening visit women who meet the inclusion/non-inclusion criteria will be offered to participate and sign the informed consent form (ICF). Initial patient's data input will be done retrospectively (case report forms [CRF] will be filled in, a patient's visit will be conducted in accordance with the routine practice and healthcare professionals (HCPs) recommendations on an individual basis). An experienced rheumatologist will collect the baseline patient's characteristics such as demographic data, clinical profile, detailed obstetric/reproductive history. Women who had pregnancies in the past will be asked about the course of all pregnancies and their outcomes. Women will be asked to provide the corresponding medical records or discharge summaries, if possible, in order to input the data from them into the CRFs (the documents will be given back to women at the same visit). The immunologic blood test will be conducted in the reference laboratory. According to clinical examination and laboratory test results (ANA, immunoassay for specific antibodies (anti-Sm, and-dsDNA), antiphospholipid antibodies (anticardiolipin antibodies, anti-β3GP1 antibodies, lupus anticoagulant, complement components C3, C4, etc.) SLE diagnosis will be made or rejected.

One follow-up visit will be conducted for those women who were referred to a laboratory testing for SLE. The visit will include the laboratory analyses assessment by an experienced rheumatologist with a subsequent confirmation or rejection of the SLE diagnosis.

The last date of enrolment - Dec 2023. Last patient last visit (approximately 4 months from the study start): patient's data input will be done for enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18-45 years old
2. Patients with reproductive issues in the past (early or late miscarriages, unexplained infertility)
3. Clinical manifestation of a suspected connective tissue disorder.
4. Women who were referred to a rheumatological settings as a part of a routine practice.
5. Provided written informed consent before any study-related procedures are performed.

Exclusion Criteria:

1. Acute infectious disease or relapse of chronic infectious disease or other condition that can affect the immunological data accuracy according to physician decision,
2. Previously confirmed by rheumatologist SLE or other immunoinflammatory disease including lupus nephritis and cutaneous or discoid lupus (acute or subacute).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study population will consist of women 18-45 years old who had reproductive issues in the past (early or late miscarriages, unexplained infertility) and were referred to a rheumatological settings as a part of a routine practice due to a suspected immunologic cause of the reproductive problems. It is estimated that approximately 2000 patients will be enrolled in approximately 15 sites in Russian Federation.
Sampling Method: Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
The frequency of confirmed SLE in women with certain clinical manifestations and reproductive issues (early or late miscarriages, unknown infertility). | Up to 5 month
  The frequency of confirmed SLE in women with certain clinical manifestations and reproductive issues (early or late miscarriages, unknown infertility).

SECONDARY OUTCOMES:
The frequency of ANA positive results in women with certain clinical manifestations and reproductive issues (early or late miscarriages, unknown infertility). | Up to 5 month
  The frequency of ANA positive results in women with certain clinical manifestations and reproductive issues (early or late miscarriages, unknown infertility).

CONTACTS AND LOCATIONS:
Locations (9):
- Russia (9):
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Orenburg
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Ufa
  - Research Site, Voronezh

REFERENCES:
- See also: D3461R00069 PRISMA Clinical Study Report (CSR) Synopsis RIMS.pdf — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3461R00069&attachmentIdentifier=2190b56a-9cc0-4d44-adc3-9aff1b5b762b&fileName=D3461R00069_PRISMA_Clinical_Study_Report_(CSR)_Synopsis_RIMS.pdf&versionIdentifier=